CLINICAL TRIAL: NCT00987324
Title: Randomized Trial of Paclitaxel-Eluting Balloon, Paclitaxel-Eluting Stent and Plain Balloon Angioplasty for Restenosis in "-Limus"-Eluting Coronary Stents
Brief Title: Efficacy Study of Paclitaxel-eluting Balloon, -Stent vs. Plain Angioplasty for Drug-eluting Stent Restenosis
Acronym: ISAR-DESIRE-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE NO. S02908
Record Dates: First submitted 2009-08-27; First posted 2009-09-30 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Heart Disease; Ischemia; Restenosis
MeSH Terms: conditions — Heart Diseases; Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paclitaxel-eluting stent (Experimental): Paclitaxel-eluting stent (Taxus)
  Interventions: Device: Taxus stent
- Plain Balloon (Active Comparator): plain balloon angioplasty
  Interventions: Device: Conventional Balloon Catheter
- Paclitaxel-eluting balloon (Experimental): SeQuent Please
  Interventions: Device: SeQuent Please

INTERVENTIONS:
Device: Taxus stent — Implantation of paclitaxel-eluting stent
  Arms: Paclitaxel-eluting stent
Device: SeQuent Please — Dilation with SeQuent Please (paclitaxel-eluting balloon)
  Arms: Paclitaxel-eluting balloon
Device: Conventional Balloon Catheter — Ryuijin, Trek
  Arms: Plain Balloon

SUMMARY:
The purpose of this randomized study is to determine which treatment option, either paclitaxel-eluting balloon, paclitaxel-eluting stent or plain balloon angioplasty is the most effective in the treatment of restenosis after implantation of "Limus"-eluting stents, (LES).

DETAILED DESCRIPTION:
The use of drug-eluting stents (DES) has led to a drastic reduction of restenosis rates compared to bare metal stents (BMS), but 5% to 10% of patients receiving DES are still in need of revascularization of the treated vessel. Two important families of drugs are used for stent coating: paclitaxel belonging to the taxane family, and the "limus"-family such as sirolimus, everolimus, zotarolimus, biolimus A9 and pimecrolimus.

Data regarding the optimal treatment of in-DES-restenosis is very limited. Implanting a new DES for in-DES-restenosis has been reported to be associated with re-restenosis rates as high as 43%. Several recent well published studies have shown a substantial reduction of restenosis using paclitaxel-eluting balloons (PEB) for de-novo lesions and BMS-restenotic lesions.

The objective of this randomized trial is to assess the hypothesis, that PEB are non-inferior to paclitaxel-eluting-stents (PES) for restenosis in "limus"-eluting-stents (LES), and both, PEB and PES, are superior to plain angioplasty in patients with restenosis after initial LES implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% restenosis after prior implantation of LES in native coronary vessels.
2. Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
3. In women with childbearing potential a negative pregnancy test is mandatory.

Exclusion Criteria:

1. Age < 18 years.
2. Cardiogenic shock.
3. Acute ST-elevation myocardial infarction within 48 hours from symptom onset.
4. Target lesion located in the left main trunk or bypass graft.
5. Target lesion located in small vessel (vessel size < 2.0 mm).
6. Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
7. Severe renal insufficiency (glomerular filtration rate ≤ 30 ml/min).
8. Contraindications to antiplatelet therapy, paclitaxel, stainless steel, cobalt, chrome.
9. Pregnancy (present, suspected or planned) or positive pregnancy test.
10. Previous enrollment in this trial.
11. Patient's inability to fully comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Percent in-segment diameter stenosis at follow-up angiography | 6-8 months

SECONDARY OUTCOMES:
In-segment minimal luminal diameter | 6-8 months
In-segment binary angiographic restenosis | 6-8 months
Combined incidence of death or myocardial infarction | 1 and 2 years
Incidence of thrombosis | 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Principal Investigator — Deutsches Herzzentrum Munich; Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum; Klaus Tiroch, MD, Study Director — Deutsches Herzzentrum
Locations (3):
- Germany (3):
  - 1. Med. Klinik, Klinikum rechts der Isar, Munich, Bavaria
  - Herz-Zentrum, Bad Krozingen
  - Deutsches Herzzentrum, Munich

REFERENCES:
- [Background] Unverdorben M, Vallbracht C, Cremers B, Heuer H, Hengstenberg C, Maikowski C, Werner GS, Antoni D, Kleber FX, Bocksch W, Leschke M, Ackermann H, Boxberger M, Speck U, Degenhardt R, Scheller B. Paclitaxel-coated balloon catheter versus paclitaxel-coated stent for the treatment of coronary in-stent restenosis. Circulation. 2009 Jun 16;119(23):2986-94. doi: 10.1161/CIRCULATIONAHA.108.839282. Epub 2009 Jun 1. PMID 19487593
- [Derived] Giacoppo D, Alvarez-Covarrubias HA, Koch T, Cassese S, Xhepa E, Kessler T, Wiebe J, Joner M, Hochholzer W, Laugwitz KL, Schunkert H, Kastrati A, Kufner S. Coronary artery restenosis treatment with plain balloon, drug-coated balloon, or drug-eluting stent: 10-year outcomes of the ISAR-DESIRE 3 trial. Eur Heart J. 2023 Apr 17;44(15):1343-1357. doi: 10.1093/eurheartj/ehad026. PMID 36807512
- [Derived] Kufner S, Cassese S, Valeskini M, Neumann FJ, Schulz-Schupke S, Hoppmann P, Fusaro M, Schunkert H, Laugwitz KL, Kastrati A, Byrne RA; ISAR-DESIRE 3 Investigators. Long-Term Efficacy and Safety of Paclitaxel-Eluting Balloon for the Treatment of Drug-Eluting Stent Restenosis: 3-Year Results of a Randomized Controlled Trial. JACC Cardiovasc Interv. 2015 Jun;8(7):877-84. doi: 10.1016/j.jcin.2015.01.031. Epub 2015 May 20. PMID 26003022
- [Derived] Byrne RA, Neumann FJ, Mehilli J, Pinieck S, Wolff B, Tiroch K, Schulz S, Fusaro M, Ott I, Ibrahim T, Hausleiter J, Valina C, Pache J, Laugwitz KL, Massberg S, Kastrati A; ISAR-DESIRE 3 investigators. Paclitaxel-eluting balloons, paclitaxel-eluting stents, and balloon angioplasty in patients with restenosis after implantation of a drug-eluting stent (ISAR-DESIRE 3): a randomised, open-label trial. Lancet. 2013 Feb 9;381(9865):461-7. doi: 10.1016/S0140-6736(12)61964-3. Epub 2012 Dec 1. PMID 23206837